CLINICAL TRIAL: NCT06734871
Title: A Clinical Study to Investigate the Safety, Efficacy, and Cellular Metabolism of CT1190B CAR-T Cell Therapy, in Patients with Relapsed/Refractory B-Cell Non-Hodgkin Lymphoma
Brief Title: A Clinical Study Exploring CT1190B in the Treatment of Patients with Relapsed/refractory B-cell Non-Hodgkin Lymphoma
Acronym: CT1190B
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aibin Liang，MD，Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Aibin Liang，MD，Ph.D., Principal Investigator, Shanghai Tongji Hospital, Tongji University School of Medicine
Organization: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT1190B-CG11001_02
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: B-Cell Non-Hodgkin Lymphoma
Keywords: CT1190B
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-T cells（ chimeric antigen receptor T cells） (Experimental): CT1190B cells infusion
  Interventions: Drug: CAR T cells

INTERVENTIONS:
Drug: CAR T cells — chimeric antigen receptor T cells

SUMMARY:
A Clinical Study to Investigate the Safety, Efficacy, and Cellular Metabolism of CT1190B CAR-T Cell therapy, in Patients with Relapsed/Refractory B-Cell Non-Hodgkin Lymphoma.

DETAILED DESCRIPTION:
This is a single-arm, open-label, dose exploratory clinical study to evaluate the safety, efficacy, cellular pharmacokinetics, and pharmacodynamics of CT1190B cells in patients with B-NHL. It is planned to enroll 6-24 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must voluntarily sign the informed consent form (ICF) and must be willing and be able to adhere to the study visit schedule and other protocol requirements and agree to be in long term follow-up (LTFU) for up to 15 years as mandated by the regulatory guidelines.
2. 18-75 years old;
3. Histologically or cytologically confirmed B-NHL;
4. Previously received at least 2 lines of systemic therapy;
5. Intolerance to last treatment, or have progressed on or after the last treatment and currently require therapy;
6. There are measurable target lesions;
7. Expected survival > 12 weeks;
8. Eastern Cooperative Oncology Group (ECOG) score 0-1;
9. Female participants of childbearing potential must have a negative pregnancy test at screening and prior to receiving preconditioning therapy and are willing to use a highly effective and reliable method of contraception for 1 year after receiving study treatment and are absolutely prohibited from donating eggs for 1 year after receiving study treatment infusion during the study; male participants are willing to use a highly effective and reliable method of contraception for 1 year after receiving study treatment if they are sexually active with a female of childbearing potential. Sperm donation is absolutely prohibited for 1 year after receiving study treatment infusions during the study for all male participants.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Has HIV, syphilis infection, active hepatitis B virus infection (HBsAg positive and HBV-DNA above the detection limit), or active hepatitis C virus infection (HCV antibody and HCV-DNA positive);
3. Has any current uncontrolled active infection, including but not limited to participants with active tuberculosis (investigator 's judgment);
4. Participants' toxicities caused by previous treatment did not recover to Common Terminology Criteria for Adverse Events (CTCAE) ≤ Grade 1, except alopecia and other events that are judged tolerable by the investigator;
5. Has received treatment for the disease within 14 days before informed consent, including but not limited to cytotoxic therapy, monoclonal antibodies or ADCs, targeted therapy, radiotherapy, epigenetic therapy, or investigational agents, or invasive investigational medical devices within 14 days before informed consent. If the radiation field covers ≤ 5% of the bone marrow reserve, the participant is eligible regardless of the end date of radiotherapy;
6. Systemic glucocorticoids equivalent to > 15 mg/day prednisone within 7 days prior to informed consent, with the exception of topical glucocorticoids;
7. Vaccination with live attenuated vaccines, inactivate vaccines or RNA vaccines within 4 weeks prior to informed consent;
8. Participants who are allergic or intolerant to preconditioning drugs, tocilizumab, or have other previous history of severe allergy such as anaphylactic shock;
9. Patients with any heart disease in the 6 months prior to screening;
10. Oxygen saturation < 92%,;
11. Presence of a second primary malignancy requiring treatment or not in complete remission within the past 2 years;
12. Major surgery within 2 weeks before informed consent or planned during the study period or within 4 weeks after giving study treatment (excluding local anesthesia such as cataract);
13. Participants are unable or unwilling to comply with the requirements of the study protocol or are otherwise unsuitable for participating in this clinical study in the investigator 's assessment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-10-13 (Estimated); Study Completion 2026-07-13 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) after CT1190B infusion | 12 months after CT1190B infusion
  An assessment of severity grade will be made according to the National Cancer Institute Common Terminology Criteria
MTD and/or dose range | Up to 28 days after CAR-T cells infusion
  Evaluate Dose limited toxicity and recommended dosage range after CT0991 infusion

SECONDARY OUTCOMES:
Overall response rate（ORR） | Evaluate at 4, 8, 12 weeks and 6,9,12month after CAR-T infusion
  The proportion of patients with complete remission （CR） /partial response (PR) after CT1190B infusion.
Complete response rate (CRR) | 12 months after CT1190B infusion
  The proportion of patients with complete response(CR) after CT1190B infusion
Duration of remission(DOR) | 12 months after CT1190B infusion
  Participants achieving CR/PR will be included in the analysis set for DOR. DOR is defined as the time from the date of confirmed response until the date of disease relapse or death from any cause, whichever occurs first.
Time to response (TTR) | 12 months after CT1190B infusion
  The time from cell infusion to the first assessment of CR or PR
Time to complete response (TTCR) | 12 months after CT1190B infusion
  The time from cell infusion to the first assessment of CR
Progression-free survival (PFS) | 12 months after CT1190B infusion
  The time from the infusion of CT1190B cells to the first assessment of disease progression or death.
Overall survival (OS) | 12 months after CT1190B infusion
  defined as the time from the date of receiving the infusion to the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Aibin Liang MD,Ph.D., Principal Investigator — Shanghai Tongji Hospital, Tongji University School of Medicine
Locations (1):
- Shanghai Tongji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No